CLINICAL TRIAL: NCT00645125
Title: A Comparative, Single-Center, Pediatric Taste Test Study of Omnicef Versus Amoxicillin Antibiotic Suspension Medications
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Angela M Nilius, PhD, Abbott
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: M02-567
Record Dates: First submitted 2008-03-22; First posted 2008-03-27 (Estimated); Last update posted 2008-03-27 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: pediatric taste test; antibiotic taste test; cefdinir; amoxicillin
MeSH Terms: interventions — Cefdinir; Amoxicillin

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: cefdinir (Omnicef)
- 2 (Active Comparator)
  Interventions: Drug: amoxicillin

INTERVENTIONS:
Drug: cefdinir (Omnicef) — 2.5 ml of strawberry cream flavored oral suspension 125 mg/5 mL
  Other Names: ABT-198; Omnicef; cefdinir
  Arms: 1
Drug: amoxicillin — 2.5 ml of bubble-gum flavored amoxicillin oral suspension 125 mg/5 mL
  Arms: 2

SUMMARY:
To compare the taste and smell acceptability scores of cefdinir (Omnicef) versus amoxicillin oral antibiotic suspension medications in pediatric subjects. It is designed to determine if Omnicef or amoxicillin is preferred to the other with regard to taste or smell.

DETAILED DESCRIPTION:
The Primary Purpose for the study is "Other". Per ClinicalTrials.gov, more information regarding the primary purpose is described here; the primary purpose for the study is to determine whether cefdinir possesses preferred taste and smell characteristics when compared to amoxicillin, a pediatric taste test.

ELIGIBILITY:
Inclusion Criteria:

* Female or male child age 4 through 8 years in good general health.
* Minimum weight of 16.3 kg (36 lb).
* Willing to comply with appropriate instructions provided to complete the study.
* Written informed consent from parent/legal guardian.

Exclusion Criteria:

* Current medical condition, that in the opinion of the Investigator or designee, could interfere with the ability to discriminate taste (e.g., common cold, sinus infection, bronchial infection, etc.).
* History of allergic reaction to cefdinir, prescription (e.g. penicillins or cephalosporins) and/or OTC medications, and/or food products.
* History of significant medical condition (e.g., GI disorders, hematological or bleeding disorders, renal or hepatic diseases).
* Use of any oral medication, vitamins or herbal supplements within 6 hours prior to tasting.
* Temperature > than 99.2°F.
* Participation in a clinical or marketing research study within the past 3 months.
* Sibling of another subject on the study, or living in the same household as another subject that has participated in a clinical or marketing research study within the past 3 months.
* Family member or close friend employed by an advertising agency, market research company and/or a company that processes or manufacturers medical or health care products.

Ages: 4 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2003-01; Primary Completion 2003-02 (Actual)

PRIMARY OUTCOMES:
Taste and smell acceptability assessment | 2 hours

SECONDARY OUTCOMES:
Adverse events assessment | 72 hours with follow-up to a satisfactory conclusion
Concomitant medications | 72 hours
Vital signs | 2 hours
Any clinically abnormal observations | 2 hours with follow-up to a satisfactory conclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Scottsdale, Arizona, United States